CLINICAL TRIAL: NCT00982566
Title: A Phase 1 Study Evaluating the Relative Oral Bioavailability of New Formulations of ABT-263 in Subjects With Cancer
Brief Title: Assess the Oral Bioavailability of a New ABT-263 Formulation in Subjects With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Mack Mabry, MD, Medical Director, Abbott
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M11-069
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2011-01

CONDITIONS: Lymphoid Malignancy; Solid Tumors
MeSH Terms: interventions — navitoclax

ARMS (16):
- Sequence I (Experimental)
  Interventions: Drug: ABT-263
- Sequence II (Experimental)
  Interventions: Drug: ABT-263
- Sequence III (Experimental)
  Interventions: Drug: ABT-263
- Sequence IV (Experimental)
  Interventions: Drug: ABT-263
- Sequence V (Experimental)
  Interventions: Drug: ABT-263
- Sequence VI (Experimental)
  Interventions: Drug: ABT-263
- Sequence VII (Experimental)
  Interventions: Drug: ABT-263
- Sequence VIII (Experimental)
  Interventions: Drug: ABT-263
- Sequence IX (Experimental)
  Interventions: Drug: ABT-263
- Sequence X (Experimental)
  Interventions: Drug: ABT-263
- Sequence XI (Experimental)
  Interventions: Drug: ABT-263
- Sequence XII (Experimental)
  Interventions: Drug: ABT-263
- Sequence XIII (Experimental)
  Interventions: Drug: ABT-263
- Sequence XIV (Experimental)
  Interventions: Drug: ABT-263
- Sequence XVI (Experimental)
  Interventions: Drug: ABT-263
- Sequence XV (Experimental)
  Interventions: Drug: ABT-263

INTERVENTIONS:
Drug: ABT-263 — Part 1: Single (oral) dose of 250 mg of Formulation B1 vs. single (oral) dose of 250 mg of Formulation A
  Arms: Sequence I; Sequence II
Drug: ABT-263 — Part 1 continued. Single (oral) dose of 250 mg of Formulation B2 vs. single (oral) dose of 250 mg of Formulation A
  Arms: Sequence III; Sequence IV
Drug: ABT-263 — Part 1: Single (oral) dose of 200 mg of Formulation C vs. single (oral) dose of 200 mg of Formulation A
  Arms: Sequence IX; Sequence V; Sequence VI; Sequence VII; Sequence VIII; Sequence X
Drug: ABT-263 — Part 1: Single (oral) dose of 200 mg of Formulation C vs. single (oral) dose of 200 mg of Formulation A
  Arms: Sequence XI; Sequence XII; Sequence XIII; Sequence XIV; Sequence XV; Sequence XVI

SUMMARY:
This is a randomized, single dose, open-label, multicenter crossover study to determine the oral bioavailability of a new ABT-263 formulation relative to that of the current ABT-263 formulation being administered in ongoing Phase 1/2a studies. Approximately 48 evaluable subjects with lymphoid malignancies, including chronic lymphocytic leukemia, and solid tumors will be enrolled in this study.

DETAILED DESCRIPTION:
Subjects who complete Part 1 of the study will be provided an opportunity to receive Formulation A under a continuous once daily dosing schedule during Part 2 of the study. Subjects enrolled in the second part of the study may continue to receive Formulation A under the continuous once daily dosing schedule for up to one year following the date of the last subject enrolled on study provided they continue to tolerate the drug, have no evidence of disease progression, and do not meet any of the protocol specific criteria for subject discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be >= 18 years of age.
2. Subject has a lymphoid malignancy (histologic or cytologic confirmation), or solid tumor (radiographic, histologic, or cytologic confirmation) that is either:

   * relapsed or refractory to standard therapy, or
   * no known effective therapy exists.
3. In the investigator's opinion, the subject's life expectancy is at least 90 days.
4. Subjects with known brain metastases must have clinically controlled neurologic symptoms, defined as surgical excision and/or radiation therapy followed by 21 days of stable neurologic function and no evidence of CNS disease progression as determined by CT or MRI within 21 days prior to the first dose of study drug.
5. If clinically indicated, subjects must have documented brain imaging (MRI or CT) negative for subdural or epidural hematoma within 28 days prior to the first dose of study drug.
6. Subject has an Eastern Cooperative Oncology Group (ECOG) performance score of <= 2.
7. Subject must have adequate bone marrow, renal and hepatic function per local laboratory reference range as follows:

   * Bone marrow: Absolute Neutrophil count (ANC) >= 1,000/µL; Platelets >= 100,000/mm3 (independent of platelet transfusions within 3 months prior to starting study drug); Hemoglobin >= 9.0 g/dL;
   * Renal function: serum creatinine <= 2.0 mg/dL or calculated creatinine clearance >= 50 mL/min;
   * Hepatic function and enzymes: AST and ALT <= 2.5 x the upper normal limit (ULN) of institution's normal range; Bilirubin <= 1.5 x ULN. Subjects with Gilbert's Syndrome may have a Bilirubin > 1.5 x ULN; Subjects with liver metastasis may have an AST and ALT of <= 5.0 x ULN;
   * Coagulation: aPTT, PT not to exceed 1.2 x ULN.
8. Female subjects must be surgically sterile, postmenopausal (for at least one year), or have negative results for a pregnancy test performed as follows:

   * At Screening on a serum sample obtained within 14 days prior to initial study drug administration, and
   * Prior to start of dosing on a urine sample if it has been > 7 days since obtaining the serum pregnancy test results.
9. Female subjects not surgically sterile or postmenopausal (for at least one year) and non-vasectomized male subjects must practice at least one of the following methods of birth control:

   * total abstinence from sexual intercourse (minimum one complete menstrual cycle prior to starting study drug);
   * a vasectomized partner;
   * hormonal contraceptives (oral, parenteral or transdermal) for at least three months prior to study drug administration;
   * double-barrier method (including condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream).
10. Subject must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

1. Subject has undergone an allogeneic stem cell transplant.
2. Subject has an underlying condition predisposing them to bleeding or currently exhibits signs of clinically significant bleeding.
3. Subject has a recent history of non-chemotherapy induced thrombocytopenic associated bleeding within one year prior to the first dose of study drug.
4. Subject has active peptic ulcer disease or other hemorrhagic esophagitis/gastritis.
5. Subject has a significant history of cardiovascular disease (e.g., MI, thrombotic or thromboembolic event in the last 6 months), renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, or hepatic disease that in the opinion of the investigator would adversely affect his/her participating in this study. Questions regarding inclusion of individual subjects should be directed to the Abbott Medical Monitor or designee.
6. Female subject is pregnant or breast-feeding.
7. Subject has a history of or an active medical condition(s) that affects absorption or motility (e.g., Crohn's disease, celiac disease, gastroparesis, short bowel syndrome, etc.).
8. Subject has tested positive for HIV (due to potential drug-drug interactions between anti retroviral inhibitors and ABT-263, as well as anticipated ABT-263 mechanism based lymphopenia that may potentially increase the risk of opportunistic infections and potential drug-drug interactions with certain anti infective agents).
9. Subject exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

   * active systemic fungal infection;
   * diagnosis of fever and neutropenia within one week prior to study drug administration.
10. Subject has received any of the following anti-cancer therapies 14 days prior to the first dose of study drug, or has not recovered to less than grade 2 clinically significant adverse effect(s)/toxicity(s) of the previous therapies:

    * chemotherapy, immunotherapy, radiotherapy;
    * hormonal therapy (with the exception of hormones for hypothyroidism or estrogen replacement therapy [ERT], or agonists required to suppress serum testosterone levels [e.g., LHRH, GnRH, etc.] for subjects with prostate cancer if on a stable dose for 21 days prior to the first dose of study drug);
    * any investigational therapy, including targeted small molecule agents
11. Subject has received a biologic agent for anti-neoplastic intent within 30 days prior to the first dose of study drug.
12. Subject is currently receiving or requires anticoagulation therapy or any drugs or herbal supplements that affect platelet function, with the exception of low-dose anticoagulation medications, such as heparin, that are used to maintain the patency of a central intravenous catheter. Note, warfarin is excluded at any dose level.
13. Subject has received aspirin within 7 days prior to the first dose of study drug and during ABT-263 administration.
14. Subject has consumed grapefruit or grapefruit products within 3 days prior to the first dose of study drug.
15. In the opinion of the investigator, the subject is an unsuitable candidate to receive ABT-263.
16. Subject has received a CYP3A inducer within 7 days prior to the first dose of study drug and during ABT-263 administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Assessment of Oral Bioavailability | Two Period and Three Period crossover design
  Assess the oral bioavailability of Formulation B1, Formulation B2, Formulation C, and Formulation D relative to that of Formulation A being assessed in ongoing Phase 1/2a ABT-263 studies

SECONDARY OUTCOMES:
Adverse Events Tabulation | Two Period and Three Period crossover design
  Safety measures include number and percentage of subjects having treatment-emergent adverse events tabulated by MedDRA system organ class and preferred term, laboratory test results, lymphocyte enumeration results, vital signs, etc.

REFERENCES:
- [Result] Xiong H, Pradhan RS, Nada A, Krivoshik AP, Holen KD, Rhodes JW, Gordon GB, Humerickhouse R, Awni WM. Studying navitoclax, a targeted anticancer drug, in healthy volunteers--ethical considerations and risk/benefit assessments and management. Anticancer Res. 2014 Jul;34(7):3739-46. PMID 24982396